CLINICAL TRIAL: NCT06377072
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of Shenqi Sherong Pill in Cervical Spondylotic Myelopathy (Qi Deficiency, Blood Stasis and Kidney Deficiency Type)
Brief Title: Efficacy and Safety of Shenqi Sherong Pill in Participants With Cervical Spondylotic Myelopathy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Hutchison Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHPL-W036-301
Record Dates: First submitted 2024-04-03; First posted 2024-04-22 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Cervical Spondylotic Myelopathy
Keywords: Qi deficiency; Blood stasis; Kidney deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shenqi Sherong Pill (Experimental): 6g per bag
  Interventions: Drug: Shenqi Sherong Pill
- Placebo (Placebo Comparator): 6g per bag
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Shenqi Sherong Pill — two bags each time, three times a day at half an hour after breakfast, lunch and dinner for 6 weeks
  Arms: Shenqi Sherong Pill
Drug: Placebo — two bags each time, three times a day at half an hour after breakfast, lunch and dinner for 6 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Shenqi Sherong Pill in participants with Mild or Moderate Cervical Spondylotic Myelopathy (qi deficiency, blood stasis and kidney deficiency type) which based on placebo-control, providing a basis for drug registration.

DETAILED DESCRIPTION:
1. Trial Design： This is a multi-center, randomized, double-blind, placebo-controlled phase III study，which plans to enroll 428 participants who will be randomized to Shenqi Sherong pill group or placebo control group. The Modified Japanese Orthopaedic Association (mJOA) Score combined with the changes of clinical symptoms and syndrome score are used as the validity index. The laboratory examination and incidence of adverse events are used as the safety index.
2. Therapeutic schedule： Participants will be provided with neck braces and recommended to wear them daily or outdoors along with health education. Participants will be treated with the investigational drug (Shenqi Sherong Pill or placebo ) by taking two bags each time, three times a day at half an hour after breakfast, lunch and dinner for 6 weeks, with a 2-week follow-up after withdrawal.

ELIGIBILITY:
Inclusion Criteria:

Participants can only be selected if they meet all the inclusion criteria

1. Age 18-75 years old (including 18 and 75 years old), gender unlimited;
2. Accord with Western medicine diagnosis standards of Cervical Spondylotic Myelopathy;
3. Accord with Chinese medicine diagnosis standards of qi deficiency, blood stasis and kidney deficiency type;
4. The disease classification was mild or moderate (13 ≤mJOA score ≤15);
5. X-ray examination of six cervical vertebrae (frontal, lateral, hyperextension and flexion lateral and double oblique) indicates cervical degenerative changes, while MRI examination indicates spinal cord compression;
6. The first diagnosis of Cervical Spondylotic Myelopathy within 3 months; for those diagnosed for more than 3 months, the investigator needs to determine that the condition is basically stable;
7. Participants voluntarily participate in this experiment and sign an informed consent.

Note: 1) CT examination is determined by the investigator according to the specific conditions of participants. 2) Imaging materials of MRI, X-ray(frontal, lateral, hyperextension and flexion and double oblique), CT examination within 3 months from the 3A Grade hospital can be accepted ; 3) If the laboratory tests and 12-lead electrocardiogram are completed in the research center on the same day before the participant signing an informed consent, the examination can not be repeated after the investigator judging.

Exclusion Criteria:

Participants should be excluded if they meet any one exclusion criteria :

1. The use of long-acting hormone drugs within 1 week before screening, or the last drug use is less than 7 half-lives, or Traditional Chinese Medicine, drugs with no marked half-life, physical therapy, etc. is less than 3 days before screening for the treatment of this disease;
2. Participants with obvious concurrent syndrome or complication (such as Hypertension after taking antihypertensive drugs who systolic pressure ≥160mmHg, or diastolic pressure ≥100mmHg , or Diabetes after taking antidiabetic drugs who fasting blood glucose ≥10.0mmol/L and so on);
3. MRI examination shows the degree of spinal stenosis is 1/2 or more, or the spinal cord compression caused by cervical spondylosis is three or more segments;
4. Participants with severe hand muscle atrophy, or spasms, or is difficult to walk independently, or urinary dysfunction;
5. Participants with cervical spine fracture, or congenital deformity of cervical spine, or ossification of ligamentum flavum, or ossification of posterior longitudinal ligament, or with neurological diseases such as lateral sclerosis and multiple sclerosis;
6. Participants with visual analogue scale(VAS) score >7 points (7 points is defined as the distance between the left end and the mark location equal to 7.0cm);
7. Participants with severe heart disease, such as myocardial infarction, unstable angina pectoris, Ⅲ to Ⅳ congestive heart failure and severe arrhythmia according to New York Heart Association (NYHA),or with severe liver and kidney diseases, or with abnormal liver and kidney function tests (Alanine aminotransferase or Aspartate aminotransferase ≥ 1.5 times the upper limit of normal, or creatinine clearance> the upper limit of normal); or with severe lung disease such as chronic bronchitis, asthma, chronic obstructive pulmonary disease(COPD) and other acute episodes;
8. Participants with cerebral infarction and serious mental disorders;
9. Woman in lactation, pregnancy, or planned pregnancy;
10. Participant is allergic constitution or known to be allergic to the components of the investigational drug;
11. Participants have participated or are participating in other clinical trials within 3 months;
12. Participants are judged unsuitable for participation by the investigators in the study.

Note: 1) If examination or efficacy index score of visit 1 and visit 2 is overlapping item, the baseline standard is based on visit 2; 2) Participant who has the abnormal laboratory examination items during screening can be arranged for retest, whether to be enrolled or not will be comprehensively evaluated by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2024-05-11 (Actual); Primary Completion 2026-01-14 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in Modified Japanese Orthopaedic Association (mJOA) score | 42±2 days
  Change in Modified Japanese Orthopaedic Association (mJOA) score (on a scale from 0 to 18, with lower scores indicating greater disability) from baseline at Day 42 after administration; the mJOA which is a clinician administered scale to evaluate four clinical dimensions; motor dysfunction score for upper and lower extremities, sensation loss and sphincter dysfunction.

SECONDARY OUTCOMES:
Change in mJOA score | 14±2 days, 28±2 days, 56±2 days
  Changes in mJOA score (on a scale from 0 to 18, with lower scores indicating greater disability) from baseline at Day 14，Day 28 and Day 56 after administration
Change in sensation of mJOA score | 14±2 days, 28±2 days, 42±2 days or 56±2 days
  Changes in sensation of mJOA score (on a scale from 0 to 3, with lower scores indicating greater disability) from baseline at Day 14, Day 28, Day 42 and Day 56 after administration
Changes in pain or stiffness score for neck and shoulder | 14±2 days, 28±2 days, 42±2 days or 56±2 days
  Changes in pain or stiffness score (on a scale from 0 to10, with higher scores indicating greater pain) for neck and shoulder from baseline at Day 14, Day 28, Day 42 and Day 56 after administration
Change in chest tightness score | 14±2 days, 28±2 days, 42±2 days or 56±2 days
  Change in chest tightness score (on a scale from 0 to10, with higher scores indicating greater tightness) from baseline at Day 14, Day 28, Day 42 and Day 56 after administration
Changes in hand and arm numbness scores | 14±2 days, 28±2 days, 42±2 days or 56±2 days
  Changes in hand and arm numbness scores (on a scale from 0 to10, with higher scores indicating greater numbness) at Day 14, Day 28, Day 42 and Day 56 after administration
Change in numbness (or pain) scores from the chest to the toes | 14±2 days, 28±2 days, 42±2 days or 56±2 days
  Changes from baseline in numbness (or pain) scores (on a scale from 0 to10, with higher scores indicating greater numbness or pain) from the chest to the toes at Day 14, Day 28, Day 42 and Day 56 after administration
Change in Motor dysfunction of the upper extremities of mJOA score | 14±2 days, 28±2 days, 42±2 days or 56±2 days
  Change in Motor dysfunction of the upper extremities of mJOA score (on a scale from 0 to 5, with lower scores indicating greater disability) at Day 14, Day 28, Day 42 and Day 56 after administration
Proportion of participants with at least 1 grade decline in Nurick grades | 14±2 days, 28±2 days, 42±2 days or 56±2 days
  Proportion of participants with at least 1 grade decline from baseline in Nurick grades (on a scale from 0 to 5, with higher scores indicating greater disability) at Day 14, Day 28, Day 42 and Day 56 after administration
Change in Traditional Chinese medicine (TCM) syndrome integrality | 14±2 days, 28±2 days, 42±2 days or 56±2 days
  Change in Traditional Chinese medicine (TCM) syndrome integrality (on a scale from 0 to 9, with higher scores indicating greater seriousness) at Day 14, Day 28, Day 42 and Day 56 after administration
Change in TCM syndrome score | 14±2 days, 28±2 days, 42±2 days or 56±2 days
  Change in TCM syndrome score (on a scale from 0 to 9, with higher scores indicating greater seriousness) at Day 14, Day 28, Day 42 and Day 56 after administration

OTHER OUTCOMES:
Serious adverse events | 14±2 days，28±2 days，42±2 days or 56±2 days
  The number and incidence of serious adverse events at Day 14, Day 28, Day 42 and Day 56 after administration
Adverse events | 14±2 days，28±2 days，42±2 days or 56±2 days
  The number and incidence of adverse events at Day 14, Day 28, Day 42 and Day 56 after administration
Vital sign (systolic and diastolic blood pressure after 10-minute rest) | 14 days before administration, 14±2 days，28±2 days，42±2 days or 56±2 days
  Number of participants with abnormal blood pressure, assessed by systolic and diastolic blood pressure before and after administration
Vital sign (body temperature) | 14 days before administration, 14±2 days，28±2 days，42±2 days or 56±2 days
  Change in body temperature from baseline or screening period at Day 14, Day 28, Day 42 and Day 56 after administration
Vital sign (respiration) | 14 days before administration, 14±2 days，28±2 days，42±2 days or 56±2 days
  Change in respiration from baseline or screening period at Day 14, Day 28, Day 42 and Day 56 after administration
Vital sign (heart rate） | 14 days before administration, 14±2 days，28±2 days，42±2 days or 56±2 days
  Change in heart rate from baseline or screening period at Day 14, Day 28, Day 42 and Day 56 after administration
Laboratory test indicator (blood routine) | 14 days before administration, 14±2 days or 42±2 days
  Number of participants with abnormal laboratory tests results, assessed by white blood cell, red blood cell, hemoglobin and platelet before and after administration
Laboratory test indicator (liver function) | 14 days before administration, 14±2 days or 42±2 days
  Number of participants with abnormal liver function, assessed by alanine aminotransferase, aspartate aminotransferase, total bilirubin, alkaline phosphatase and gamma-glutamyl transpeptidase before and after administration
Laboratory test indicator (kidney function) | 14 days before administration, 14±2 days or 42±2 days
  Number of participants with abnormal kidney function, assessed by serum creatinine, urinary microalbumin, urinary albumin to creatinine ratio, urinary N-Acetyl-β-D-glucosaminidase and urinary creatinine before and after administration
Laboratory test indicator (fasting glucose) | 14 days before administration, 14±2 days or 42±2 days
  Change in fasting glucose before and after administration
Laboratory test indicator (urine routine and urinary sediment count) | 14 days before administration, 14±2 days or 42±2 days
  Number of participants with abnormal urine analysis, assessed by urinary white blood cell, urinary red blood cell, urinary protein and urinary proportion before and after administration
Laboratory test indicator (stool routine and occult blood) | 14 days before administration, 14±2 days or 42±2 days
  Number of participants with abnormal stool analysis, assessed by stool routine and occult blood before and after administration
Electrocardiogram(ECG) QT Interval | 14 days before administration, 14±2 days or 42±2 days
  Change in ECG QT Interval before and after administration
ECG QTc Interval | 14 days before administration, 14±2 days or 42±2 days
  Change in ECG QTc Interval before and after administration
ECG QRS Interval | 14 days before administration, 14±2 days or 42±2 days
  Change in ECG QRS Interval and PR Interval before and after administration
ECG PR Interval | 14 days before administration, 14±2 days or 42±2 days
  Change in ECG PR Interval before and after administration
Pathological sign (Hoffmann sign) | 14 days before administration, 14±2 days, 28±2 days, 42±2 days or 56±2 days
  Changes of Hoffmann sign from baseline or screening period at Day 14, Day 28, Day 42 and Day 56 after administration
Pathological sign (Babinski sign) | 14 days before administration, 14±2 days, 28±2 days, 42±2 days or 56±2 days
  Changes of Babinski sign from baseline or screening period at Day 14, Day 28, Day 42 and Day 56 after administration
Concomitant medication | 14 days before administration, 14±2 days, 28±2 days, 42±2 days or 56±2 days
  Number of participants with concomitant medication throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: Bolai Chen, doctor, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China